CLINICAL TRIAL: NCT06635954
Title: A Prospective Real World Evidence Study (PROWES) for Concordance Rate of Blood-based 3D Genome Conformation Mapping (Episwitch CiRT®) to Identify Likelihood of Response and Actual Response Rates to PD-(L)-1 Checkpoint Inhibitors Across Multiple Oncological Indications.
Acronym: PROWES
Status: Recruiting | Type: Observational
Sponsor: Oxford Biodynamics Inc. (Industry)
Collaborators: Community Clinical Oncology Research Network, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: OB202401
Record Dates: First submitted 2024-09-05; First posted 2024-10-10 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-10

CONDITIONS: Cancer; Immunotherapy; PD-1; PD-L1; Immune Checkpoint Therapy
Keywords: immunotherapy; immune checkpoint inhibitor; ICI therapy; ICI; Immune Checkpoint Inhibitor therapy; Episwitch; Episwitch CiRT; Immune Related Adverse Event; IRAE; cancer; PD-1; PD-L1
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this research is to test whether a blood-based 3D genome conformation mapping test called the Episwitch CiRT® can help to identify likelihood of response to PD-(L)-1 checkpoint inhibitors (a class of cancer drugs) across multiple oncological indications by comparing the results to actual treatment responses for cancer patients.

DETAILED DESCRIPTION:
The Episwitch CiRT® (Checkpoint inhibitor Response Test) predicts how a patient will respond to immune checkpoint inhibitor (ICI) therapies by delivering a binary response likelihood profile (High Probability vs. Low Probability).

Patients who have been diagnosed with stage III and IV cancer and who are candidates and/or planned to receive immune check point inhibitors as a therapy now or in near future will be offered the Episwitch CiRT™ before starting treatment or if on active treatment. Those patients with high probability of response to ICI will undergo repeat testing every three months. Patients will be followed for up to six months. Treatment administered, disease-free survival, overall survival, stable disease, progressive disease, complete response, time to recurrence, physician questionnaires and patient-reported outcomes will be recorded for six months. Comprehensive data of Social Determinants of Health (SDoH) will be collected to identify any correlation to unmet Health Related Social Needs (HrSN) and likelihood to response and/or resistance

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Stage III or IV cancer
3. Selected by their healthcare provider to receive the Episwitch CiRT® test according to the current evidence-based schedule (per protocol) as part of their standard of practice.
4. ECOG performance status ≤ 2
5. Clinically eligible for ICI therapy
6. Able to read, understand and provide written informed consent.
7. Willing and able to comply with the study requirements

Exclusion Criteria:

1. Pregnant or breastfeeding
2. History of bone marrow or organ transplant
3. Contra indication for receiving Immune Check Point inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a stage III or IV cancer diagnosis that have been identified and indicated by their healthcare provider to receive immune check point inhibitors as a therapy now or in the near future.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2026-05-14 (Estimated); Study Completion 2027-05-14 (Estimated)

PRIMARY OUTCOMES:
Correlation between low probability of response prediction and actual response rate to Immune Checkpoint Inhibitor Therapy | From enrollment to the final Episwitch test at week 24
  At the time of enrollment, case report forms will be completed that capture the patient's current and previous treatments, stage of disease, and prognosis. After receiving results from Episwitch CiRT, a follow up case report form will be completed that captures the response prediction from the test as well as the patient's response to their current treatment, and whether or not that treatment is an ICI therapy. The patients on ICI that receive results that indicate low probability of response will be compared to their actual response to treatment.
Establish Health Economics Outcomes Research based on the potential cost savings from foregoing ICI therapy based on Episwitch CiRT prediction of response | From time of enrollment to the 24-week follow up test results
  Patients that are predicted to have a low probability of response to ICI therapy and are receiving ICI therapy will be identified throughout the study via case report forms. We will estimate drug cost savings based on the amount of ICI therapy received by the patient. We will also capture any immune related adverse events from the ICI therapy and account for any costs related to these reactions. This will all be used as a rough model and predictor of the potential cost savings of using the Episwitch CiRT in treatment decisions.
Determine the existence of a correlation between Social Determinants of Health and test results and patient outcomes | From time of enrollment to the 24-week follow up test results
  Upon enrollment, patients will complete a Social Determinants of Health Questionnaire that captures the following information: ethnicity, race, quality of housing, housing insecurity, highest education, employment status, insurance, income, how frequently patients talk to those they care about, transportation needs, refugee status, and lack of access to the following resources food, utilities, phone, clothing, childcare, and medicine/health care.
  The responses will be used to identify patients that have no, low, or high needs and compare these groups' testing results and outcomes to each other. Further or more in-depth analysis may be needed to understand correlations between SDOH and ICI therapy outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Mathis, MD, Study Director — Oxford BioDynamics
Locations (3):
- United States (3):
  - Eastern Connecticut Hematology and Oncology, Norwich, Connecticut
  - Cancer Center of Middle Georgia, Dublin, Georgia
  - Carolina Blood and Cancer Care Associates, Rock Hill, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided
This topic has not been discussed in depth between us and the sponsor. The priority now is to recruit and collect data to show the efficacy of this test. Please reach out to Joseph DeSimone or Ryan Mathis if more information is desired.

REFERENCES:
- See also: What is CiRT? — https://mycirt.com/index.html?utm_medium=email-signature%20&utm_campaign=cirt-video#video_20692
- See also: Oxford Biodynamics — https://www.oxfordbiodynamics.com/
- See also: Community Clinical Oncology Research Network (CCORN) — https://www.ccorn.net/